CLINICAL TRIAL: NCT02954939
Title: The Effect of Mycophenolate Mofetil and Cyclophosphamide on the Lymphocyte Subsets and Relationship With Relapse
Brief Title: The Effect of Mycophenolate Mofetil and Cyclophosphamide on the Lymphocyte Subsets in Patients With Proliferative Lupus Nephritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: UW12-389
Record Dates: First submitted 2016-09-13; First posted 2016-11-04 (Estimated); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Lupus Nephritis
Keywords: lupus nephritis; lymphocyte subsets; cytokines; mycophenolate mofetil; cyclophosphamide
MeSH Terms: conditions — Lupus Nephritis | interventions — prednylidene

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MMF-MMF (Active Comparator): Class III/IV+V LN patients who receive prednisolone (PRED) (0.8mg/kg/d) plus mycophenolate mofetil (MMF) (1g bd) as induction-maintenance therapy
  Interventions: Drug: MMF-MMF
- CTX-AZA (Placebo Comparator): Class III/IV+V LN patients who receive prednisolone (PRED) (0.8mg/kg/d) plus Cyclophosphamide (CTX) (1.5-2mg/kg/d) followed by Azathioprine (AZA) (1-1.5mg/kg/d) as induction-maintenance therapy
  Interventions: Drug: CTX-AZA

INTERVENTIONS:
Drug: MMF-MMF — Class III/IV+/-V lupus nephritis patients to receive PRED+MMF
  Other Names: PRED; MMF
  Arms: MMF-MMF
Drug: CTX-AZA — Class III/IV+/-V lupus nephritis patients to receive PRED+CTX followed by AZA
  Other Names: PRED; CTX; AZA
  Arms: CTX-AZA

SUMMARY:
This study investigated the effect of mycophenolate mofetil and cyclosphosphamide on lymphocyte subsets in patients with proliferative lupus nephritis. Patients with biopsy-proven Class III/IV+/-V LN were randomized to received: 1) prednisolone (0.8mg/kg/day) plus CTX (1.5-2mg/kg/d) for 6 months) followed by Azathioprine (AZA) (1-1.5mg/kg/d) maintenance; OR 2) prednisolone (0.8mg/kg/d) plus MMF (1g bd) for 6 months, followed by MMF (tapered according to clinical status) as maintenance. The lymphocyte subsets and serum cytokine profiles will be measured at 4-, 12-, and 24-, 36- and 48 weeks after induction treatment. The lymphocyte subsets and serum cytokine profiles will be compared between the two treatment regimens, and also correlated with subsequent risk of relapse.

DETAILED DESCRIPTION:
This study investigated the effect of mycophenolate mofetil and cyclosphosphamide on lymphocyte subsets in patients with proliferative lupus nephritis. Patients with biopsy-proven Class III/IV+/-V LN were randomized to received: 1) prednisolone (0.8mg/kg/day) plus CTX (1.5-2mg/kg/d) for 6 months) followed by Azathioprine (AZA) (1-1.5mg/kg/d) maintenance; OR 2) prednisolone (0.8mg/kg/d) plus MMF (1g bd) for 6 months, followed by MMF (tapered according to clinical status) as maintenance. The lymphocyte subsets and serum cytokine profiles will be measured at 4-, 12-, and 24-, 36- and 48 weeks after induction treatment. The lymphocyte subsets and serum cytokine profiles will be compared between the two treatment regimens, and also correlated with subsequent risk of relapse.

ELIGIBILITY:
Inclusion Criteria:

- 1. Patients with biopsy proven Class III/IV+/-V LN (ISN/RPS classification) and active nephritis as indicated by an increase of proteinuria >1g/day and/or rise in serum creatinine by >15% compared with baseline, with or without serological reactivation.

2. Willing to give informed consent

Exclusion Criteria:

1. Patients who have received calcineurin inhibitors or proliferation signal inhibitors as maintenance immunosuppression in the preceding 3 months
2. Patients have received biologics therapy (e.g. rituximab, abatacept) in the preceding 12 months
3. Patients who are pregnant or lactating

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Lymphocyte subset profile (CD8+ T cells, CD4+ Th1, Th2, Th17 & Treg), Naïve & memory B cells, plasma cells | 48 weeks

SECONDARY OUTCOMES:
serum cytokine profile (IL-2, IL-5, IL-6, IL-7, IL-10, IL-17, IL-21, IL-23, IFN-alpha, IFN-gamma, TGF-beta) | 48 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong